CLINICAL TRIAL: NCT04349033
Title: Virtual Human Technology for Patients With Chronic Pain: Experimental Study of Pain Neuroscience and Emotional Disclosure
Brief Title: Virtual Human Technology for Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, Mark A. Lumley, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UP-19-00230
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Chronic Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Emotional Disclosure and Brain Education (Experimental): Patients are interviewed about stress and other emotional issues and are educated about how emotions and the brain influence pain.
  Interventions: Behavioral: Emotional Disclosure and Brain Education
- Emotional Disclosure only (Active Comparator): Patients are interviewed about stress and other emotional issues only.
  Interventions: Behavioral: Emotional Disclosure Only
- Pain Information Control (Placebo Comparator): Patients are interviewed about their pain history and experience.
  Interventions: Behavioral: Pain Information Control

INTERVENTIONS:
Behavioral: Emotional Disclosure and Brain Education — Patients are interviewed about a number of aspects of their lives (stress, other illnesses, personality, adverse childhood experiences), and these are explored as part of education of the brain's role in their pain.
  Arms: Emotional Disclosure and Brain Education
Behavioral: Emotional Disclosure Only — Patients are interviewed about a number of aspects of their lives, but without brain education
  Arms: Emotional Disclosure only
Behavioral: Pain Information Control — Patients are interviewed about their pain history and other basic, non-disclosure information about their health.
  Arms: Pain Information Control

SUMMARY:
The experimental study compares three virtual human interviews of patients with chronic musculoskeletal pain: Emotional disclosure and brain, emotional disclosure only, basic information control. Effects on attitudes and clinical outcomes at 1-month follow-up are assessed.

DETAILED DESCRIPTION:
Emotional disclosure about stressors and other private experiences has been found to be helpful for some people with chronic musculoskeletal pain. Also, helping patients understand the role of the brain in pain has been helpful. We have developed a virtual human interviewer to help patients talk about their pain and their lives. We will conduct an experimental study to compare the effects of several different types of VH interviews. Patients with chronic pain will be randomized to receive one of three VH interviews: emotional disclosure and brain education; emotional disclosure alone; or a control basic pain interview. Patients will be assessed at baseline and 1-month follow-up on a range of attitudinal and clinical measures to determine how these different interviews affect outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic musculoskeletal Pain

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doerte U Junghaenel, PhD, Principal Investigator — University of Southern California; Mark A Lumley, PhD, Principal Investigator — Wayne State University
Locations (1):
- University of Southern California Center for Self-report Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Full, anonymized data set
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 1 year after study end, for 5 years.
Access Criteria: Contact the study PI

REFERENCES:
- [Derived] Junghaenel DU, Schneider S, Lucas G, Boberg J, Weinstein FM, Richeimer SH, Stone AA, Lumley MA. Virtual Human-Delivered Interviews for Patients With Chronic Pain: Feasibility, Acceptability, and a Pilot Randomized Trial of Standard Medical, Psychosocial, and Educational Interviews. Psychosom Med. 2023 Sep 1;85(7):627-638. doi: 10.1097/PSY.0000000000001228. Epub 2023 Jun 16. PMID 37363989

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started on February 10, 2021, and the study concluded on August 1, 2021
Groups:
- Emotional Disclosure and Brain Education ("Educational Interview"): Patients are interviewed about stress and other emotional issues and are educated about how emotions and the brain influence pain.
  Emotional Disclosure and Brain Education: Patients are interviewed about a number of aspects of their lives (stress, other illnesses, personality, adverse childhood experiences), and these are explored as part of education of the brain's role in their pain.
- Emotional Disclosure Only ("Psychosocial Interview"): Patients are interviewed about stress, psychosocial risk factors, and other emotional issues, but with no feedback or brain-related education.
  Emotional Disclosure Only: Patients are interviewed about a number of aspects of their lives, but without brain education
- Pain Information Control ("Standard Interview"): Patients are interviewed about their pain history and experience.
  Pain Information Control: Patients are interviewed about their pain history and other basic, non-disclosure information about their health.
Period: Overall Study
Arm/Group | Emotional Disclosure and Brain Education ("Educational Interview") | Emotional Disclosure Only ("Psychosocial Interview") | Pain Information Control ("Standard Interview")
Started | 29 | 34 | 31
Completed | 26 | 33 | 30
Not Completed | 3 | 1 | 1
Not completed — Lost to Follow-up | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Emotional Disclosure Only ("Psychosocial Interview"): Patients are interviewed about stress and other emotional issues only.
  Emotional Disclosure Only: Patients are interviewed about a number of aspects of their lives, but without brain education
- Total: Total of all reporting groups
Arm/Group | Emotional Disclosure and Brain Education ("Educational Interview") | Emotional Disclosure Only ("Psychosocial Interview") | Pain Information Control ("Standard Interview") | Total
Number analyzed (Participants) | 29 | 34 | 31 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.03 (14.99) | 56.65 (13.68) | 45.84 (13.21) | 51.04 (14.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 28 | 82
  Male | 3 | 6 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 1 | 1 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 22 | 30 | 24 | 76
  More than one race | 2 | 1 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 34 | 31 | 94

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: Brief Pain Inventory (average of the 4 pain intensity rating items: highest, lowest, average, now). Range: 0.0 to 10.0 (higher = more severe pain)
Time Frame: Change from Baseline to 1-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Emotional Disclosure and Brain Education ("Educational Interview") | Emotional Disclosure Only ("Psychosocial Interview") | Pain Information Control ("Standard Interview")
Number analyzed (Participants) | 29 | 34 | 31
score on a scale | -0.21 (0.19) | -0.56 (0.17) | -0.09 (0.17)

2. Secondary Outcome: Pain Interference
Description: Brief Pain Inventory (7 interference items; range: 0.0 to 10.0; higher = more interference)
Time Frame: Change from Baseline to 1-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Emotional Disclosure and Brain Education ("Educational Interview") | Emotional Disclosure Only ("Psychosocial Interview") | Pain Information Control ("Standard Interview")
Number analyzed (Participants) | 29 | 34 | 31
score on a scale | -0.82 (0.37) | -1.27 (0.33) | -0.31 (0.35)

3. Secondary Outcome: Pain Stages of Change Questionnaire
Description: Pain Stages of Change Questionnaire assesses readiness / motivation to engage in pain self-management. Sum of subscales of Contemplation + Action + Maintenance - Precontemplation; Range = 0 to 12; higher scores = more readiness to change
Time Frame: Change from Baseline to 1-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Emotional Disclosure and Brain Education ("Educational Interview") | Emotional Disclosure Only ("Psychosocial Interview") | Pain Information Control ("Standard Interview")
Number analyzed (Participants) | 29 | 34 | 31
score on a scale | 0.30 (0.26) | -0.18 (0.23) | -0.30 (0.24)

4. Secondary Outcome: Pain Catastrophizing Scale
Description: Pain catastrophizing (range: 0.0 to 4.0; higher scores = more catastrophizing)
Time Frame: Change from Baseline to 1-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Emotional Disclosure and Brain Education ("Educational Interview") | Emotional Disclosure Only ("Psychosocial Interview") | Pain Information Control ("Standard Interview")
Number analyzed (Participants) | 29 | 34 | 31
score on a scale | -0.19 (0.11) | -0.15 (0.10) | -0.06 (0.10)

5. Secondary Outcome: Emotional Distress
Description: Self-rating of how "depressed," "anxious," "angry," and "guilty" participant was during last week on 0 to 4 scale. Ratings averaged; higher means = more distress
Time Frame: Change from Baseline to 1-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Emotional Disclosure and Brain Education ("Educational Interview") | Emotional Disclosure Only ("Psychosocial Interview") | Pain Information Control ("Standard Interview")
Number analyzed (Participants) | 29 | 34 | 31
score on a scale | -0.31 (0.14) | -0.16 (0.13) | -0.06 (0.13)

ADVERSE EVENTS:
Time Frame: During the 1-hour virtual interview with the patients, which was held remotely (via telehealth) with a research assistant, and then during the 1-month follow-up period, through the completion of on-line questionnaires.
Arm/Group | Emotional Disclosure and Brain Education ("Educational Interview") | Emotional Disclosure Only ("Psychosocial Interview") | Pain Information Control ("Standard Interview")
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/34 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/34 | 0/31
Other Adverse Events (participants affected / at risk) | 0/29 | 0/34 | 0/31

LIMITATIONS AND CAVEATS:
Patient debriefing was conducted at the end of the VH session and before the follow-up assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT04349033/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT04349033/SAP_001.pdf